CLINICAL TRIAL: NCT05620745
Title: Resilience as a Mediator Between Adverse Life Events and Emotional Behavioral Problems in Children and Adolescents and Comparison Between Individuals With Attention-Deficit /Hyperactive Disorder and Controls
Brief Title: Comparison of Resilience Between ADHD and Controls.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMRPG3M1351
Record Dates: First submitted 2022-10-26; First posted 2022-11-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-10

CONDITIONS: ADHD; Resilience; Stress
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To explore if resilience serves as a mediator between adverse life events and emotional and behavioral problems, and compare the difference of resilience and its mediating effects between children and adolescents with and without ADHD.

ELIGIBILITY:
Inclusion Criteria:

* ADHD; Control without ADHD

Exclusion Criteria:

* ASD, other major physical and psychiatric diseases

Ages: 6 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: cases ever diagnosed as ADHD; Controls who didn't recieve ADHD diganosis before.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
comparison of resilience between ADHD and controls | up to 1 month
  We will use SPSS and SPSS PROCESS to analyze the data. The t-test will be used to compare the difference of resilience performance between child and adolescents with and without ADHD.
  Pearson correlation analyses will be adopted to calculate the relationships between all variables.
  Moreover, the bias-corrected method was used to estimate the 95% bootstrap confidence interval (CI)of the mediating and moderating effects of resilience between adverse life events and emotional and behavioral problems. Finally, we would compare if there is difference between the mediating effect of resilience in group with ADHD and control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung memorial hospital, Taoyuan, Taiwan